CLINICAL TRIAL: NCT03358524
Title: Effects of Vitamin E (Alfa-Tocoferol) Supplementation on Isoprostane and Lipid Profile of Obese Adolescent in Jakarta, Indonesia
Brief Title: Effects of Vitamin E Supplementation on Free Radicals and Fat Level of Obese Adolescence in Jakarta, Indonesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ali Alhadar, Pediatric Fellowship at Pediatric Nutrition and Metabolic disease, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Obesity, Adolescent; Oxidative Stress
MeSH Terms: conditions — Pediatric Obesity | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin E 400 IU (Experimental): Vitamin-E Capsule (alpha-tocopherol) 400 IU once per day orally for 8 weeks
  Interventions: Drug: Vitamin E 400 UNT
- Placebo (Placebo Comparator): Placebo capsule once per day orally for 8 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Vitamin E 400 UNT — Vitamin-E capsule (alpha tocopherol) 400 IU (once per day)
  Other Names: Vitamin E
  Arms: Vitamin E 400 IU
Drug: Placebo oral capsule — sugar capsule manufactured to mimic vitamin E capsule once per day
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study evaluate supplementation of vitamin E (alpha-tocopherol) in obese adolescent. Half of the patient will receive vitamin E and the other half received placebo

DETAILED DESCRIPTION:
One of obesity treatments that play important role is antioxidant diet. The effects of vitamin E supplementation as an antioxidant treatment in obese adolescent have not been concluded yet in Indonesia. The primary aim of this study is to observe oxidative stress biomarker (isoprostane) in obese teenagers who consume vitamin E for 2 months. The secondary aim is to observe their body mass index and lipid profile after supplementation

The study is randomized, double blind, placebo controlled trial in design and employed a consecutive sampling technique to sample subjects of 70 obese adolescent age 14 - 18 in senior high schools Jakarta.

Blood tests of lipid profile (total cholesterol, HDL, LDL, Triglyceride), fasting blood glucose, liver function (AST,ALT) and oxidative stress biomarker (isoprostane) were taken for every subject after done fasting for 12 hours.

This study is a randomized allocation and double blind technique. subjects divided into two groups, which one group receiving treatment of vitamin E and other group receiving placebo.

The dose and duration of vitamin E treatment is 400 IU per day for 2 months. At the end of treatment, all subjects had to run the same medical interview, physical examination and blood test.

ELIGIBILITY:
Inclusion Criteria:

* Obesity BMI ≥ p95 (CDC growth curve)

Exclusion Criteria:

* Consuming antioxidants drug regularly within recruiting time
* Consuming Orlistat

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Isoprostane (oxidative stress) | 8 weeks
  pg/ml

SECONDARY OUTCOMES:
Total Cholesterol | 8 weeks
  mg/dl
LDL Cholesterol | 8 weeks
  mg/dl
HDL Cholesterol | 8 weeks
  mg/dl
Triglycerides | 8 weeks
  mg/dl
Body weight | 8 weeks
  kilograms
Body Height | 8 weeks
  centimeters
BMI | 8 weeks
  kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- SMA Labschool, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided